CLINICAL TRIAL: NCT05768048
Title: SMA Natural History Study Evaluating Long Term Trajectories of SMA Patients Receiving or Not Disease-modifying Treatments
Brief Title: Long Term Trajectories of SMA Patients Receiving or Not Disease-modifying Treatments
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: University of Milan (Other); Bambino Gesù Hospital and Research Institute (Other); University of Messina (Other); Gaslini Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 4863
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational multicenter retrospective and prospective study on natural history of SMA also considering the 'new natural history' secondary to the availability of commercially available therapies.

All the patients enrolled to date in the Italian registry, if not part of clinical trials, will be included in the present study.

DETAILED DESCRIPTION:
This is an observational multicenter retrospective and prospective study on natural history of SMA also considering the 'new natural history' secondary to the availability of commercially available therapies.

All patients affected by Spinal Muscular Atrophy 5q, irrespective of genotype, phenotype, age, treatment status or gender will be enrolled in the study .

The study aims to i) better understand the natural history of the disease in untreated patients in terms of functional aspects, concomitant illnesses, quality of life ii) describe the patterns of disease progression in treated and untreated patients in terms of functional aspects, concomitant illnesses, quality of life iii) Describe all the patients treated with the available therapies in Italy, in terms of demographic (age, location etc..) and epidemiological data All data from patients included in the study will be collected at each visit, following the clinical care protocols of each centre. Following care recommendation patients are generally routinely assessed at least every 6 months and, in many cases, every 4 months.

We plan to obtain

* Longitudinal changes in untreated patients: The possibility to access reliable retrospective data will provide the opportunity to record long term functional data in untreated patients.
* Yearly analysis of longitudinal changes in treated patients:
* Two-year results of the validation of new measures (SMA HI, SMAIS): reporting the validation process (inter- and intra-observer reliability, internal consistency) and changes in relation to functional measures

ELIGIBILITY:
Inclusion Criteria:

all patients with mutationsin the SMAN1 gene

Exclusion Criteria:

unable to proviude consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients affected by Spinal Muscular Atrophy 5q, irrespective of genotype, phenotype, age, treatment status or gender
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2027-11-27 (Estimated); Study Completion 2027-11-27 (Estimated)

PRIMARY OUTCOMES:
motor function using the HFMSE (min score 0, max 74 indicating best performance) | 5 years
  motor scale

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Istituto Gaslini, Genova
  - Nemo Sud, Messina
  - Centro Clinico nemo, Milan
  - Ospedale Bambino gesu, Rome
  - Policlinico gemelli, Rome

IPD SHARING:
Plan to Share IPD: No
only aggregate data are allowed from consent